CLINICAL TRIAL: NCT01976390
Title: A Prospective, Randomized, Single Center Pilot Study Comparing Patient and Graft Survival, Adverse Events and Tolerability of Zortress® (Everolimus) Versus Rapamune® (Sirolimus) in Combination With Low Dose Neoral® (Cyclosporine) Dosed by C2 Monitoring, in Deceased and Living Donor Renal Transplant Recipients Under a Thymoglobulin® (Antithymocyte Globulin) and Rapid Steroid Induction Protocol.
Brief Title: Comparing Everolimus and Sirolimus in Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2013H0229
Record Dates: First submitted 2013-10-20; First posted 2013-11-05 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2021-11

CONDITIONS: Renal Failure
Keywords: Kidney; Kidney transplant; Renal failure; End Stage Renal Disease; kidney transplant recipient
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic | interventions — Everolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zortress (Everolimus) (Active Comparator): Zortress will be started on day of transplant and initially dosed at 0.75 mg twice a day (12 hours apart) dosed simultaneously with Neoral.
  Interventions: Drug: Everolimus
- Rapamune (Sirolimus) (Active Comparator): Rapamune will be dosed on day of transplant at 5 mg/d, decreasing to 3 mg/d.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Everolimus — 0.75mg twice a day, Orally, starting on day of transplant
  Other Names: Zortress
  Arms: Zortress (Everolimus)
Drug: Sirolimus — 5mg, Orally, starting on day of transplant; decreasing to 3mg
  Other Names: Rapamune
  Arms: Rapamune (Sirolimus)

SUMMARY:
This study is being done to compare the effectiveness and safety of two different kidney transplant immunosuppression drugs, Zortress (the study drug) and Rapamune (which is used in the current standard immunosuppression regimen).

DETAILED DESCRIPTION:
Zortress is FDA approved, is used as standard of care at some other institutions, and may also be given as standard of care if it is believed to be the best immunosuppression regimen for a particular kidney transplant recipient. The rationale for testing Zortress vs. Rapamune is to determine which of these drugs is more effective in preventing chronic rejection of the transplanted kidney. Because these two drugs are related to each other there is no current literature addressing the replacement of Rapamune with Zortress in an immunosuppression regimen, therefore the goal of this study is to compare these two immunosuppression drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent before any assessment is performed.
2. Primary renal transplant recipients between ages 18 and 75 years of age.
3. Females capable of becoming pregnant must have a negative pregnancy test prior to transplantation and practice an effective form of birth control for the duration of the study and 12 weeks after discontinuation of the study drug if applicable.

Exclusion Criteria:

1. Total cholesterol > 300 mg/dl or triglycerides > 400 mg/dl despite lipid lowering therapy
2. Pre-existing bone marrow suppression (White Blood Cell count of < 3000, platelets < 100,000)
3. Active infection (Hepatitis B Virus, HIV)
4. Malignancy (except for adequately treated squamous or basal cell skin carcinoma) unless patient has written clearance from an Oncologist or if patient has had no malignancy for at least 2 years prior to the transplant
5. Allergy or intolerance to Zortress, Rapamune, cyclosporine, or Anti-thymocyte globulin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amer Rajab, MD, Principal Investigator — OSU Wexner Medical Center
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zortress (Everolimus) | Rapamune (Sirolimus)
Started | 41 | 19
Completed | 41 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Kidney Transplant Patients at Ohio State University Medical Center taking either everolimus or sirolimus.
Groups:
- Total: Total of all reporting groups
Arm/Group | Zortress (Everolimus) | Rapamune (Sirolimus) | Total
Number analyzed (Participants) | 41 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.9) | 49.5 (12.2) | 49.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 22
  Male | 24 | 14 | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Endpoint of Graft Survival (Non-death Censored) and Biopsy Proven Acute Rejection at 1 Year
Description: The primary objective of this pilot study will be to determine equivalency of Zortress® as compared to Rapamune® when used in our de novo immunosuppression regimen following renal transplantation. The primary endpoint will be a composite endpoint of graft survival (non-death censored) and biopsy proven acute rejection at 1 year. The primary outcome of immunosuppressive protection would be studied in our Thymoglobulin and rapid steroid discontinuation protocol, with "half-dose" Neoral as described above.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Zortress (Everolimus) | Rapamune (Sirolimus)
Number analyzed (Participants) | 41 | 19
Participants
  graft survival (non-death censored) at 1 year | 40 | 19
  biopsy proven acute rejection at 1 year | 38 | 19

ADVERSE EVENTS:
Time Frame: 1 year
Description: Electronic medical records
Arm/Group | Zortress (Everolimus) | Rapamune (Sirolimus)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/19
Serious Adverse Events (participants affected / at risk) | 35/41 | 17/19
Other Adverse Events (participants affected / at risk) | 0/41 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zortress (Everolimus) (N=41) | Rapamune (Sirolimus) (N=19)
Serious Adverse Effects (General disorders) | 35 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2013-05-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT01976390/Prot_SAP_000.pdf
  • Informed Consent Form (2012-02-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT01976390/ICF_001.pdf